CLINICAL TRIAL: NCT04940689
Title: Opioid-Free Anesthesia in Cardiac Surgery
Acronym: OFACS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/0399/HP
Record Dates: First submitted 2021-05-07; First posted 2021-06-25 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Lidocaine; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard arm (Active Comparator): General anesthesia strategy with morphine:
  * Within 10 minutes before the induction of general anesthesia: administration of a placebo of 50 mL of 0.9% NaCl by slow IV
  * The anesthetic induction will be carried out by an intravenous hypnotic (propofol or etomidate) combined with IV curare and remifentanil (morphine derivative) IV for a concentration target of 4 ng / mL.
  * Maintenance of anesthesia will be carried out with propofol or a halogenated gas (sevoflurane or desflurane) in continuous administration (qs bispectral index 40-60) and remifentanil (target concentration 1-10 ng / mL). The administration of curare will be carried out as needed. In order to anticipate the sudden end of the analgesia, an administration of morphine 0.15 mg / kg IV will be carried out 30 minutes before the end of the intervention as recommended
  Interventions: Drug: Remifentanil
- OFA arm (Experimental): General anesthesia strategy without morphine
  * Within 10 minutes before the induction of general anesthesia: pre-induction dose of dexmedetomidine 0.5 g / kg and lidocaine 1.5 mg / kg by slow IV.
  * The anesthetic induction will be carried out by an intravenous hypnotic (propofol or etomidate) combined with an IV curare
  * The maintenance of the anesthesia will be carried out by propofol or a halogenated gas (sevoflurane or desflurane) in continuous administration (qsp bispectral index 40-60), dexmedetomidine 0.5-1.0 g / kg / h, lidocaine 2 mg / kg / h. The administration of curare will be carried out as needed.
  Interventions: Drug: Dexmédétomidine 0.5 g/kg + lidocaine 1.5 mg/kg

INTERVENTIONS:
Drug: Dexmédétomidine 0.5 g/kg + lidocaine 1.5 mg/kg — The patient will be anesthetized with Dexmedetomidine 0.5 g / kg + lidocaine 1.5 mg / kg for the induction instead of morphin.
  Other Names: experimental
  Arms: OFA arm
Drug: Remifentanil — The patient will be anesthetized with morphin.
  Other Names: Control
  Arms: Standard arm

SUMMARY:
The use of morphine derivatives is widespread for performing general anesthesia. However, opioids have their own side effects: respiratory depression, digestive ileus, cognitive dysfunction, postoperative hyperalgesia, nausea-vomiting or even negative effects on inflammation or adrenal function. The advent of new molecules, with analgesic properties that do not pass through opioid receptors, has allowed the emergence of the concept of anesthesia without morphine (opioid free anesthesia OFA). These molecules are essentially: dexmedetomidine, ketamine, lidocaine. Thus, the use of ketamine is currently recommended in the event of major surgery in order to limit postoperative pain and hyperalgesia. Likewise, the use of dexmedetomidine in place of an opioid during bariatric surgeries has been shown to reduce postoperative pain and intraoperative hemodynamic manifestations. In addition, it would also reduce the incidence of postoperative cognitive dysfunction. A recent meta-analysis even suggested a decrease in length of stay, mechanical ventilation, atrial fibrillation and mortality with the use of dexmedetomidine in the perioperative period. The combined use of various non-morphine analgesic molecules therefore opens the way to anesthesia without morphine, and a French multicenter study on this strategy in general non-cardiac surgery is currently underway. Cardiac surgery is characterized by significant postoperative pain, a high incidence of cognitive dysfunction, and frequent and sometimes significant respiratory complications. An OFA strategy could therefore be beneficial to these patients, but no study has yet addressed the subject.

DETAILED DESCRIPTION:
The objective of our work is therefore to assess the beneficial effects of OFA versus strategy with intraoperative opioids on postoperative complications related to opioids.

ELIGIBILITY:
Inclusion Criteria:

* Patients having planned cardiac surgery under cardiopulmonary bypass, with at least one coronary artery bypass grafting and rf at least one internal mammary artery as graft; possible association with aortic valve replacement
* Patient having red and understood the information letter and signed the consent form
* For women : of childbearing age, need to confirm the absence of an active pregnancy by a negative blood pregnancy test within 48 hours prior to inclusion / menopausal (amenorrhea not medically induced for at least 12 months before the inclusion visit)
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Preoperative treatment with morphine or its derivatives (including tramadol) in the 15 days preceding the inclusion visit
* Pre-existing high-degree conduction disorder
* Bradycardia < 50 bpm
* Oxygen therapy prior to inclusion
* Heart failure with LVEF <40%
* BMI ≥ 35 kg/m²
* Myocardial suffering in the 5 days preceding inclusion
* Patient in shock
* Known adrenal insufficiency and / or long-term systemic corticosteroid treatment (equivalent to hydrocortisone hemisuccinate ≥ 20 mg / day)
* Combined surgery other than aortic valve
* Long-term non-invasive ventilation (including for obstructive sleep apnea syndrome)
* Any antecedent or active practice (s) of drug addiction;
* Contraindication to one of the experimental and / or non-experimental treatments: dexmedetomidine, lidocaine, dexamethasone, ketamine, remifentanil or morphine
* Acute cerebrovascular pathology,
* Severe hepatic insufficiency (factor V level <50%),
* Pre-existing cognitive disorders,
* Patient for whom the CAM-ICU questionnaire cannot be carried out (deaf patients for example),
* Pregnant or parturient or breastfeeding woman
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection / under guardianship or guardianship
* Patient participating in another drug trial or having participated in another drug trial within 1 month before randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
To assess the impact of general anesthesia strategy without the use of opioids (OFA) on the incidence of major postoperative complications related to opioids compared to the reference strategy using opioids. | 48 hours post-surgery
  Composite criterion consisting of the appearance 48 hours after the surgery of an intestinal ileus, and / or of an alteration of the neurological state, and / or of an acute respiratory failure, and / or of a death

SECONDARY OUTCOMES:
To assess the impact of OFA on the incidence of postoperative nausea and vomiting. | 48 hours post-surgery
  Existence of post-surgery nausea
To assess the impact of OFA on the incidence of postsurgery pain. | 48 hours post-surgery
  Number of post-surgery pain episodes at rest (VAS ≥ 3) and total morphine consumption
To assess the impact of OFA on the incidence of atrial rhythm disturbances and / or ventricular postsurgery shock states. | 48 hours post-surgery
  Appearance of non-preexisting atrial fibrillation and/or of postsurgery ventricular rhythm disturbances and/or high degree cardiac conduction disorders
To assess the impact of OFA on the incidence of acute post-surgery renal failure, | 48 hours post-surgery
  Onset of acute renal failure defined by a KDIGO score ≥ 1
To assess the impact of the OFA on the incidence of post-surgery adrenal insufficiency, | 24 hours post-surgery
  Incidence of relative adrenal insufficiency 24 hours postoperatively by performing a synacthene test. An increase in cortisol levels <250 nmol / L within one hour of the injection of 250 µg of tetracosactide is a diagnosis
Evaluate the impact of the OFA on the impact of the length of ICU and hospital stay Evaluate the impact of the OFA on the impact of the length of post-surgeryhospital stay | Within 2 months after surgery
  Number of days in the hospital
Evaluate the impact of the OFA on the incidence of postoperative mortality | Within 2 months after surgery
  Number of deaths
Persistence of chronic pain evaluated during a telephone call | 3 months after surgery
  simple numerical scale, from 0 to 10
Persistence of chronic pain evaluated during a telephone call | 3 months after surgery
  neuropatic pain questionnaire (DN4), from 0 to 10
To assess the impact of OFA on the incidence of shock | 48 hours post-surgery
  Presence of cardiogenic shock and vasoplegic syndrome
To assess the myocardial pain | 48 hours post-surgery
  maximum troponin plasma level
To assess the intraoperative safety | intraoperative periode
  Existence of bradycardia requiring atropine adminitsrtation and/or appearance of arterial hypotension or hypertension

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Rouen University Hospital, Rouen, France, Normandy
  - Amiens Univesrity Hospital, Amiens
  - CAEN university Hospital, Caen
  - Lille Hopistal University, Lille
  - Montpellier University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Yes
Data generated by this trial will not be publicly available but upon reasonable request to the corresponding author (Emmanuel Besnier, emmanuel.besnier@chu-rouen.fr). In this case, data will be totally deidentified. Requesters should provide a structured and detailed protocol for the proposed study and the reasons for reusing data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From results publication to 10 years

REFERENCES:
- [Derived] Besnier E, Moussa MD, Thill C, Vallin F, Donnadieu N, Ruault S, Lorne E, Scherrer V, Lanoiselee J, Lefebvre T, Sentenac P, Abou-Arab O. Opioid-free anaesthesia with dexmedetomidine and lidocaine versus remifentanil-based anaesthesia in cardiac surgery: study protocol of a French randomised, multicentre and single-blinded OFACS trial. BMJ Open. 2024 Jun 3;14(6):e079984. doi: 10.1136/bmjopen-2023-079984. PMID 38830745